CLINICAL TRIAL: NCT00306462
Title: Randomized Double-Blinded Trial of Magnesium Sulfate Tocolysis Versus Nifedipine Tocolysis in Women With Preterm Labor Between 24 to 32 6/7 Weeks' Gestation
Brief Title: Trial of Magnesium Sulfate Tocolysis Versus Nifedipine Tocolysis in Women With Preterm Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment in past year, lack of interest
Sponsor: University of Cincinnati (Other)
Collaborators: University Hospital (Other)
Responsible Party: Baha Sibai, MD/Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-12-27-01
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Premature Birth; Premature Labor
Keywords: Premature Labor; Premature Birth; Magnesium sulfate; Nifedipine
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Magnesium Sulfate; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Intravenous magnesium sulfate or placebo
  Interventions: Drug: Magnesium sulfate
- 2 (Active Comparator): Oral nifedipine or placebo
  Interventions: Drug: Oral Nifedipine or placebo

INTERVENTIONS:
Drug: Magnesium sulfate — Intravenous magnesium sulfate 6g bolus, then increased by 1 g/hour till a maximum of 5g/hour; gradually wean down to 2 g/hour for a total of 48 hours once uterine contractions is < 6/hour.
  Arms: 1
Drug: Oral Nifedipine or placebo — Oral nifedipine or placebo at 20 mg every 30 minutes for the first hour, then 20 mg every 3 to 6 hours not to exceed 180 mg in 24 hours, keep maintenance dose at 20 mg every 3 to 6 hours for a total of 48 hours if uterine contractions is < 6/hour.
  Other Names: Oral procardia
  Arms: 2

SUMMARY:
Primary Hypothesis:

Acute tocolysis (48 hours) using oral nifedipine is more effective than intravenous magnesium sulfate in prolonging pregnancy in women with preterm labor with intact membranes between 24 and 32 6/7 weeks' gestation.

DETAILED DESCRIPTION:
Primary Objective:

To compare the efficacy of oral nifedipine versus IV magnesium sulfate on the rate of preterm delivery at <37 weeks in women with preterm labor between 24 and 32 6/7 weeks gestation.

Secondary Objective:

1. To compare maternal side effects between the two tocolytic agents
2. To compare neonatal morbidities between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Women in preterm labor between 24 to 32 6/7 weeks' gestation with intact membranes with an age range of 15 to 50 years old.

Exclusion Criteria:

* Cervical dilatation of ≥ 6 cm
* Maternal contraindication to tocolysis
* Known fetal anomalies
* Suspected chorioamnionitis
* Nonreassuring fetal heart tracing
* Vaginal bleeding due to placenta previa or abruptio placenta
* Preterm premature rupture of membranes
* Prolapsed membranes
* Human immunodeficiency virus positive
* Multiple gestation
* Patients on procardia within 24 hours of po intake
* Magnesium sulfate tocolysis prior to randomization
* Patient refusal

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Delivery <37 weeks' gestation, Delivery <34 weeks' gestation, Delivery <32 weeks' gestation | 4 years

SECONDARY OUTCOMES:
Maternal complications associated with each drugs. Neonatal morbidities associated with prematurity | 4 years and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Baha Sibai, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Crowley P. Prophylactic corticosteroids for preterm birth. Cochrane Database Syst Rev. 2000;(2):CD000065. doi: 10.1002/14651858.CD000065. PMID 10796110
- [Background] Crowther CA, Hiller JE, Doyle LW. Magnesium sulphate for preventing preterm birth in threatened preterm labour. Cochrane Database Syst Rev. 2002;(4):CD001060. doi: 10.1002/14651858.CD001060. PMID 12519550
- [Background] Huddleston JF, Sanchez-Ramos L, Huddleston KW. Acute management of preterm labor. Clin Perinatol. 2003 Dec;30(4):803-24, vii. doi: 10.1016/s0095-5108(03)00114-3. PMID 14714923
- [Background] King JF, Flenady VJ, Papatsonis DN, Dekker GA, Carbonne B. Calcium channel blockers for inhibiting preterm labour. Cochrane Database Syst Rev. 2003;(1):CD002255. doi: 10.1002/14651858.CD002255. PMID 12535434
- [Background] Morales WJ, Madhav H. Efficacy and safety of indomethacin compared with magnesium sulfate in the management of preterm labor: a randomized study. Am J Obstet Gynecol. 1993 Jul;169(1):97-102. doi: 10.1016/0002-9378(93)90138-9. PMID 8333483
- [Background] Papatsonis DN, Kok JH, van Geijn HP, Bleker OP, Ader HJ, Dekker GA. Neonatal effects of nifedipine and ritodrine for preterm labor. Obstet Gynecol. 2000 Apr;95(4):477-81. doi: 10.1016/s0029-7844(99)00596-7. PMID 10725475
- [Background] Ramsey PS, Rouse DJ. Magnesium sulfate as a tocolytic agent. Semin Perinatol. 2001 Aug;25(4):236-47. doi: 10.1053/sper.2001.27546. PMID 11561911
- [Result] Glock JL, Morales WJ. Efficacy and safety of nifedipine versus magnesium sulfate in the management of preterm labor: a randomized study. Am J Obstet Gynecol. 1993 Oct;169(4):960-4. doi: 10.1016/0002-9378(93)90035-h. PMID 8238157
- [Result] Haghighi L. Prevention of preterm delivery: nifedipine or magnesium sulfate. Int J Gynaecol Obstet. 1999 Sep;66(3):297-8. doi: 10.1016/s0020-7292(99)00095-8. PMID 10580682
- [Result] Larmon JE, Ross BS, May WL, Dickerson GA, Fischer RG, Morrison JC. Oral nicardipine versus intravenous magnesium sulfate for the treatment of preterm labor. Am J Obstet Gynecol. 1999 Dec;181(6):1432-7. doi: 10.1016/s0002-9378(99)70388-1. PMID 10601925
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046